CLINICAL TRIAL: NCT07146997
Title: Evaluation of Combined Effect of Oral Premedications on Enhancing the Effectiveness of Inferior Alveolar Nerve Block in Mandibular Teeth With Symptomatic Irreversible Pulpitis
Brief Title: Evaluating the Combined Effect of Oral Premedications on Inferior Alveolar Nerve Block Effectiveness
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Zahoor khan (Other)
Collaborators: HITEC-Institute of Medical Sciences (Other)
Responsible Party: Sponsor-Investigator, Zahoor khan, Dr Zahoor khan BDS FCPS, HITEC-Institute of Medical Sciences
Organization: HITEC-Institute of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: Dental/HITEC/IRB/60
Record Dates: First submitted 2025-08-13; First posted 2025-08-28 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2023-11

CONDITIONS: Symptomatic Irreversible Pulpitis
MeSH Terms: interventions — Sugars; Ibuprofen; serratiopeptidase

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group I - Placebo Group (Control) (Placebo Comparator): Group I - Placebo:
  Participants will receive an oral placebo capsule identical in appearance to the active medications, administered one hour before IANB, to serve as the control group for comparison of anesthetic effectiveness
  Interventions: Dietary Supplement: Patients in this group will receive an oral placebo (e.g., sugar tablet or inert capsule) 1 hour before the IANB
- Group II - Ibuprofen Group (Active Comparator): Group II - Ibuprofen:
  Participants will receive a single oral dose of ibuprofen (400 mg) administered one hour prior to IANB to evaluate its effect on improving anesthetic success in symptomatic irreversible pulpitis
  Interventions: Drug: Patients will receive ibuprofen (400-600 mg, standard therapeutic dose) orally, 1 hour prior to IANB
- Group III - Serratiopeptidase Group (Active Comparator): Group III - Serratiopeptidase:
  Participants will receive a single oral dose of serratiopeptidase (10 mg) one hour before IANB to assess its effect on enhancing anesthetic efficacy in symptomatic irreversible pulpitis
  Interventions: Drug: Group III - Serratiopeptidase Group
- Group IV - Combination Group (Ibuprofen and Serratiopeptidase) (Active Comparator): Group IV - Combination (Ibuprofen and Serratiopeptidase):
  Participants will receive a single oral dose of ibuprofen (400 mg) and serratiopeptidase (10 mg) one hour before IANB to assess the combined effect on enhancing anesthetic success in symptomatic irreversible pulpitis
  Interventions: Combination Product: Group IV - Combination Group (Ibuprofen and Serratiopeptidase)

INTERVENTIONS:
Dietary Supplement: Patients in this group will receive an oral placebo (e.g., sugar tablet or inert capsule) 1 hour before the IANB — Group I - Placebo Group (Control) Intervention: Patients in this group will receive an oral placebo (e.g., sugar tablet or inert capsule) 1 hour before the IANB.
  Purpose: This group serves as the control to establish a baseline anesthetic success rate without active premedication.
  Expected Outcome: Lower IANB success rate due to lack of anti-inflammatory intervention.
  Arms: Group I - Placebo Group (Control)
Drug: Patients will receive ibuprofen (400-600 mg, standard therapeutic dose) orally, 1 hour prior to IANB — Group II - Ibuprofen Group Intervention: Patients will receive ibuprofen (400-600 mg, standard therapeutic dose) orally, 1 hour prior to IANB.
  Purpose: Ibuprofen is a nonsteroidal anti-inflammatory drug (NSAID) that inhibits COX-1 and COX-2 enzymes, reducing prostaglandin synthesis and inflammation, which can enhance anesthetic efficacy.
  Expected Outcome: Improved IANB success rate compared to placebo, but possibly lower than combination therapy.
  Arms: Group II - Ibuprofen Group
Drug: Group III - Serratiopeptidase Group — Group III - Serratiopeptidase Group Intervention: Patients will receive serratiopeptidase (10 mg or standard dose) orally, 1 hour before the IANB.
  Purpose: Serratiopeptidase is a proteolytic enzyme with anti-inflammatory, mucolytic, and fibrinolytic properties. It helps reduce tissue inflammation by breaking down inflammatory mediators and possibly inhibiting prostaglandin production.
  Expected Outcome: Improved IANB success rate compared to placebo; effectiveness may vary compared to ibuprofen alone
  Arms: Group III - Serratiopeptidase Group
Combination Product: Group IV - Combination Group (Ibuprofen and Serratiopeptidase) — Group IV - Combination Group (Ibuprofen and Serratiopeptidase) Intervention: Patients will receive a combination of ibuprofen and serratiopeptidase orally, 1 hour before IANB. The doses will be the same as those used in Groups II and III, respectively.
  Purpose: This group is designed to test the synergistic effect of combining an NSAID (ibuprofen) and a proteolytic enzyme (serratiopeptidase) to maximize inflammation control and increase the success of IANB in inflamed pulp tissue.
  Expected Outcome: Highest success rate of IANB due to dual action on prostaglandin inhibition and tissue inflammation reduction
  Arms: Group IV - Combination Group (Ibuprofen and Serratiopeptidase)

SUMMARY:
This clinical study investigates whether the combination of ibuprofen and serratiopeptidase as oral premedication can enhance the effectiveness of the inferior alveolar nerve block (IANB) in patients with symptomatic irreversible pulpitis in mandibular teeth. Due to the inflammatory nature of the condition, standard IANB often fails, possibly due to prostaglandin-induced nerve sensitization.

A total of 96 patients meeting specific inclusion criteria will be divided into four groups:

Placebo

Ibuprofen alone

Serratiopeptidase alone

Combination of ibuprofen and serratiopeptidase

Pain levels will be measured using the Verbal Numerical Scale (VNS) at various treatment stages. The success of anesthesia will be determined by the absence or presence of pain during access cavity preparation and initial root canal instrumentation. Statistical analysis will compare the effectiveness between groups, with the goal of determining whether combined premedication significantly improves IANB success.

The study is conducted at the Department of Operative Dentistry & Endodontics, HITEC-IMS Taxila, over a period of six months.

DETAILED DESCRIPTION:
Detailed Description of the Study Title Evaluation of Combined Effect of Oral Premedication on Enhancing the Effectiveness of Inferior Alveolar Nerve Block in Mandibular Teeth with Symptomatic Irreversible Pulpitis

Background and Rationale Achieving effective local anesthesia is a cornerstone of pain-free endodontic treatment. The inferior alveolar nerve block (IANB) is commonly used to anesthetize mandibular teeth. However, its success rate significantly drops in cases of symptomatic irreversible pulpitis, primarily due to inflammatory changes, nerve sensitization, and increased prostaglandin production. Prostaglandins, synthesized via the cyclooxygenase (COX-1 and COX-2) pathway, lower the pain threshold and reduce anesthetic efficacy.

Nonsteroidal anti-inflammatory drugs (NSAIDs) like ibuprofen are widely used to reduce inflammation by inhibiting COX enzymes, thereby decreasing prostaglandin production. Several studies have shown that preoperative ibuprofen can enhance the effectiveness of IANB. However, other studies report conflicting results.

On the other hand, serratiopeptidase is a proteolytic enzyme known for its anti-inflammatory, mucolytic, fibrinolytic, and analgesic properties. It also acts on the COX pathway and reduces prostaglandin levels, offering a potentially synergistic effect with NSAIDs.

This study aims to evaluate the combined effect of ibuprofen and serratiopeptidase as premedication on improving the effectiveness of IANB in mandibular teeth with symptomatic irreversible pulpitis. To date, no published research has explored the combined preoperative use of these two agents for this purpose.

Objective To evaluate whether combined oral premedication with ibuprofen and serratiopeptidase enhances the anesthetic effectiveness of inferior alveolar nerve block in mandibular teeth diagnosed with symptomatic irreversible pulpitis, compared to individual or no premedication.

Research Question Does the combined oral premedication of ibuprofen and serratiopeptidase improve the success rate of IANB more than when either drug is used alone or a placebo is given?

Hypothesis Null Hypothesis (H₀): Combined oral premedication with ibuprofen and serratiopeptidase has no significant effect on the effectiveness of IANB.

Alternative Hypothesis (H₁): Combined oral premedication with ibuprofen and serratiopeptidase enhances the effectiveness of IANB.

Study Design A prospective, randomized, controlled clinical trial using non-probability consecutive sampling.

Study Setting and Duration Conducted in the Department of Operative Dentistry & Endodontics, Dental College HITEC-IMS, Taxila, over a period of 6 months following ethical and institutional approval.

Sample Size A total of 96 patients will be enrolled (24 patients per group), calculated using 80% study power, a 5% level of significance, and expected success rates of ibuprofen (78%) and serratiopeptidase (76.3%).

Eligibility Criteria

Inclusion Criteria:

Age between 18-45 years

Mandibular molars or premolars with deep carious lesions

Clinical diagnosis of symptomatic irreversible pulpitis

Normal periodontal ligament (PDL) space on IOPA

No analgesics taken within 12 hours of treatment

Exclusion Criteria:

Presence of periapical radiolucency

Teeth tender to percussion

Allergy to any of the drugs or anesthetic solution

Pregnancy or systemic illness

Failure of local anesthesia on first attempt

Patients not providing informed consent

Group Allocation

Patients will be randomly assigned to one of four groups:

Group Premedication Dosage (to be specified) I Placebo - II Ibuprofen [Standard dose] III Serratiopeptidase [Standard dose] IV Ibuprofen + Serratiopeptidase [Standard dose each]

Methodology

After obtaining informed consent, patients will receive their assigned premedication orally one hour prior to anesthesia. Pain levels will be assessed using the Verbal Numerical Scale (VNS) at the following stages:

Before premedication

After IANB administration

During access cavity preparation

At first file placement in the canal

The IANB will be performed using 2% lidocaine with 1:100,000 epinephrine (MEDICAINE - Korea). Lip numbness will confirm successful anesthesia. If lip numbness is absent, supplemental anesthesia will be administered. Only those achieving effective block (confirmed lip numbness) will proceed to treatment.

Pain perception will be categorized:

0-3: No or mild pain (Success)

4-10: Moderate to severe pain (Failure)

Rubber dam isolation and root canal procedures will be done by a single operator to ensure consistency. Data will be recorded in a coded proforma (Annexure B).

Data Collection Tools Patient data will be collected using a structured proforma (Annexure B).

Consent forms will be signed in both English and Urdu (Annexure A).

Data Analysis

Data will be analyzed using SPSS version 26:

Quantitative variables (age, weight): Mean ± Standard Deviation

Qualitative variables (gender, group success rates): Frequencies and Percentages

Statistical Tests:

Chi-square test for qualitative comparisons

Post hoc Bonferroni test for intergroup pain score comparisons

P-value ≤ 0.05 will be considered statistically significant

Ethical Considerations Approval will be obtained from the CPSP registration and research cell and the Institutional Review and Ethical Board.

All participants will be informed in detail and will sign a bilingual consent form.

Confidentiality of patient data will be strictly maintained.

Participation is voluntary, and patients may withdraw at any time.

Expected Outcome It is anticipated that patients receiving combined ibuprofen and serratiopeptidase premedication will show a higher success rate of IANB compared to those receiving either drug alone or placebo. If confirmed, this approach could improve anesthetic protocols in endodontic treatment of inflamed mandibular teeth.

ELIGIBILITY:
* Inclusion criteria:

  * Age group of subjects between 18-45 years
  * Normal PDL appearance on IOPA
  * No analgesics taken 12 hours prior to study
  * Mandibular molars and premolars with deep carious lesion having sign and symptom of symptomatic irreversible pulpitis
* Exclusion criteria:

  * Presence of periapical radiolucency on IOPA
  * Teeth tender to percussion /traumatic teeth
  * Allergy to medications/anesthetic solution
  * Pregnant patient & systemic illness
  * Patient in which local anesthesia is not effective in first attempt
  * Patient not giving consent

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2023-11-23 (Actual); Primary Completion 2024-11-23 (Actual); Study Completion 2024-11-23 (Actual)

PRIMARY OUTCOMES:
Effectiveness of Inferior Alveolar Nerve Block (IANB | Time Frame: Perioperative
  Effectiveness of Inferior Alveolar Nerve Block (IANB)
  Measured by the success rate of IANB in mandibular teeth with symptomatic irreversible pulpitis.
  Success is defined as:
  No pain or mild pain (VNS score 0-3) during:
  Access cavity preparation
  First file placement in the root canal
  Failure is defined as:
  Moderate to severe pain (VNS score 4-10) during the same stages.
  This will be compared among the four study groups (Placebo, Ibuprofen, Serratiopeptidase, and Combination therapy).

CONTACTS AND LOCATIONS:
Overall Officials: Dr Zahoor Dr Zahoor khan, BDS, FCPS, Principal Investigator — Dental college HITEC-IMS Taxila
Locations (1):
- HITEC-IMS Taxila, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: As my study has not been published yet. so i have provided the related parent articleIn link above URL section just for reference & support of the study — https://pubmed.ncbi.nlm.nih.gov/33548329/